CLINICAL TRIAL: NCT07322588
Title: Enhancing Medication for Opioid Use Disorder Retention With Post-Release Contingency Management
Brief Title: Reentry Incentives and Support for Engagement With Contingency Management
Acronym: RISE-CM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Clatsop Behavioral Healthcare (Unknown); Oregon Health Authority (Other); Clatsop County Corrections (Unknown)
Responsible Party: Principal Investigator, Linda Peng, Assistant Professor of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028902; Agreement #184714 (Other Grant/Funding Number: Oregon Health Authority)
Record Dates: First submitted 2025-12-01; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
Keywords: contingency management; opioid use disorder; incarceration; reentry
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Palliative Care; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RISE-CM Intervention (Other): All participants are enrolled in the intervention arm.
  Interventions: Other: Reentry Incentives and Support for Engagement with Contingency Management (RISE-CM) Intervention

INTERVENTIONS:
Other: Reentry Incentives and Support for Engagement with Contingency Management (RISE-CM) Intervention — Participants receive gift card rewards for attending MOUD appointments and counseling appointments after release from incarceration.

SUMMARY:
People leaving jail face a very high risk of overdose, especially in the first few weeks after release. Staying on medication for opioid use disorder (MOUD) can greatly reduce this risk, but many people stop treatment during this transition. This study is testing whether a program that offers rewards, called contingency management (CM), can help people stay on MOUD after they return to the community.

In this study, people who are taking MOUD in jail can choose to participate. While still incarcerated, they complete one visit where they may receive a small incentive, such as commissary credit or snacks, for enrolling in the CM program. After they leave jail, participants can earn gift cards when they attend their MOUD appointments and counseling sessions.

Participants may take part in the study for up to three months after release. During this time, they can earn up to $600 in incentives based on their treatment engagement. Researchers will also ask participants to complete a baseline survey and a survey at 3 months. We will also review medical records to confirm whether they continued their MOUD.

The researchers want to learn whether this adapted contingency management program is feasible, acceptable to participants, and helpful for supporting treatment engagement after release from jail. The findings will help determine whether this approach should be tested in a larger study to reduce overdose risk and improve health during the post-release period.

ELIGIBILITY:
Inclusion Criteria:

* Be adults (age ≥18 years) currently incarcerated at Clatsop County Jail
* Be enrolled in the jail's MOUD program at the time of recruitment
* Plan to continue MOUD with Clatsop Behavioral Healthcare upon release
* Speak English and be able to provide informed consent

Exclusion Criteria

Exclusion Criteria:

* Are unable to provide informed consent due to cognitive impairment or acute psychiatric instability
* Are scheduled for transfer to a different facility or geographic location that prevents post-release participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving medication for opioid use disorder | 1, 2, and 3 months
  We will assess patient reported receipt of medication for opioid use disorder and also use chart review to determine whether patients are receiving medications and three different time points.

SECONDARY OUTCOMES:
Number of contingency management sessions attended | 3 months
  Number of contingency management sessions attended per participant
Total contingency management rewards earned | 3 months
  Total dollar amount of contingency management rewards earned by participant throughout the intervention
Addiction Severity | Baseline and 3 months
  Participant reported addiction severity using the validated Brief Addiction Monitor, a 17-item, multidimensional progress monitoring tool designed to support the provision of measurement-based care to patients commencing and matriculating through treatment for substance use disorders (SUD). The BAM items assess: (1) Risk for relapse or worsening severity of SUD (Range 0-180 with higher scores indicating higher risk), (2) Protective behaviors that support recovery and resistance to relapse (Range 0-180 with higher score indicating higher protective factors), and (3) Use of alcohol and other substances (Range 0-90 with higher score indicating higher substance use).
Recovery Capital | Baseline and 3 months
  Participant reported survey on recovery capital using the validated "Brief Assessment of Recovery Capital (BARC-10)" survey. Score range 10-60 with higher scores indicating higher recovery capital.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Peng, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Clatsop County Corrections, Warrenton, Oregon, United States

IPD SHARING:
Plan to Share IPD: No